CLINICAL TRIAL: NCT02858921
Title: A Phase II, Randomised, Open Label Study of Neoadjuvant Dabrafenib, Trametinib and / or Pembrolizumab in BRAF V600 Mutant Resectable Stage IIIB/C Melanoma
Brief Title: Neoadjuvant Dabrafenib, Trametinib and/or Pembrolizumab in BRAF Mutant Resectable Stage III Melanoma
Acronym: Neo Trio
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Melanoma Institute Australia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIA2015/179
Record Dates: First submitted 2016-07-16; First posted 2016-08-08 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Melanoma
Keywords: Neoadjuvant Therapy; Pembrolizumab; Dabrafenib; Trametinib; Pathological response; RECIST; Immune response; BRAF; Randomised; Stage IIIB/C; Biomarkers, Tumour; Biomarkers, Drug response; Metabolic Response
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — dabrafenib; trametinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sequential D + T, THEN Pembrolizumab (Experimental): Dabrafenib 150mg orally twice a day + Trametinib 2mg orally once a day for 1 week, then followed by treatment with Pembrolizumab 2mg/kg delivered intravenously at weeks 1, 3, and 6, then once every 3 weeks from week 6 for 46 weeks.
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Drug: Pembrolizumab
- Concurrent D + T AND Pembrolizumab (Experimental): Dabrafenib 150mg orally twice a day + Trametinib 2mg orally once a day + Pembrolizumab 200mg intravenously once every 3 weeks for 6 weeks, the Pembrolizumab alone for 46 weeks
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Drug: Pembrolizumab
- Pembrolizumab ONLY (Experimental): Pembrolizumab 200mg intravenously once every 3 weeks alone for 52 weeks.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Dabrafenib — Dabrafenib, a 4-(3-aminosulfonylphenyl)-5-(pyrimidine-3-yl) thiazole, is a potent and selective inhibitor of B-RAF kinase activity with a mode of action consistent with adenosine triphosphate (ATP)-competitive inhibition, and is approved as monotherapy in BRAF V600E-mutant advanced/metastatic melanoma.
  Other Names: Tafinlar
  Arms: Concurrent D + T AND Pembrolizumab; Sequential D + T, THEN Pembrolizumab
Drug: Trametinib — Trametinib, a pyrido - pyrimidine derivative, is a potent and highly selective allosteric non-competitive inhibitor of MEK1/MEK2 activation and kinase activity has been approved as monotherapy in BRAF (V600E)-mutant and BRAF (V600K)-mutant melanoma.
  Other Names: Mekinist
  Arms: Concurrent D + T AND Pembrolizumab; Sequential D + T, THEN Pembrolizumab
Drug: Pembrolizumab — Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2.
  Other Names: Keytruda

SUMMARY:
This study aims to determine which of 3 drug combinations best reduces the size of tumour prior to surgery for advanced melanoma and prevents the recurrence of melanoma after surgery.

DETAILED DESCRIPTION:
The new drug options for advanced melanoma include oncogene-targeted therapy (such as dabrafenib, trametinib and vemurafenib) and immune checkpoint blockade (such as pembrolizumab, nivolumab and ipilimumab). These drugs have shown remarkable efficacy and have regulatory approval for metastatic disease. However, most patients with advanced disease eventually progress. It is unknown if earlier treatment with systemic therapy after surgery improves long term survival or what is the optimal sequencing or combination of therapy. An efficient method of assessing drugs and combinations in humans is critical, particularly as combinations of molecularly targeted and/or immune therapies may have similar signals for efficacy in pre-clinical models, and recapitulation of the human immune system in animal models is limited.

Neoadjuvant clinical trials in patients with resectable but bulky stage III/IV melanoma allows for the rapid evaluation of drug activity in humans utilising multiple clinical endpoints (metabolic response with Positron Emission Tomography [PET], clinical response with Computed Tomography [CT] imaging, pathological response, relapse-free survival and overall survival) and translational endpoints (morphological, genetic and immunophenotyping of tumour and blood).

Surgery remains the standard of care for resectable Stage III or IV melanoma, despite the recent drug therapy advances described above. The Food and Drug Administration (FDA) has recently expanded the approved use of ipilimumab to include a new use as adjuvant therapy for patients with resectable stage III / IV melanoma, to lower the risk of relapse following surgery. Neoadjuvant therapy in this group of patients may also result in improved survival rates and in the duration of local and distant disease control, with reduced surgical morbidity and the potential for early elimination of microscopic metastatic disease.

There is an emerging and rapidly growing evidence base of the value of combining targeted and immunotherapies in a number of histological subtypes of cancers. The support for a potential synergy between the two treatment modalities has been established, as has the increased toxicity profile. Both single agent BRAF inhibitors and combined BRAF and MEK inhibitors induce a marked clonal T cell infiltrate in responding melanoma metastases early during treatment (day 7-15), which is transient, and is not present at progression. Concurrently, melanoma tumour antigen and the programmed death-ligand 1 (PDL1) expression increase early during treatment.

It is unknown whether there is potential for converting a subset of patients who fail either immunotherapy or targeted therapy alone into long-term responders by treating with programmed cell death protein 1 (PD-1) inhibitors in conjunction with mitogen-activated protein kinases (MAPK) targeted therapies. Furthermore, it is unclear whether the PD-1 inhibitor would be best combined sequentially or concurrently with MAPK inhibitors. Mouse models have provided a clear rational for combining these treatments upfront, however there is no human tissue evidence to guide best combination strategies.

The question of how best to maximize clinical outcome via concurrent versus sequential targeted and immune therapy may be explored efficiently in the human neoadjuvant setting, with detailed interrogation of multiple biopsies early during treatment. Immunological, proteomic and genetic features in tissue and blood provide an in vivo assessment of tumour responsiveness to therapy. This may enable more selective application of therapeutic agents to patients who are more likely to benefit. Such findings would improve the therapeutic index and cost effectiveness of these agents. Earlier systemic therapy prior to surgery also means earlier targeting of distant micrometastases that could become the source of future disease relapse.

The rationale for this study design is therefore based on the hypothesis that one week of targeted therapy may be sufficient to induce an enhanced tumoral immunity to result in a higher pathological and clinical response using the 'Response Evaluation Criteria In Solid Tumors' (RECIST) guidelines when followed sequentially with pembrolizumab, than either pembrolizumab alone or the combination of targeted therapy and pembrolizumab upfront.

The potential for toxicities that could affect adherence to the combined study treatments are recognised, as additive, overlapping or unforeseen adverse events may occur with the triple combination. The adverse event profiles and safety-related interruption to treatment will therefore be assessed in conjunction with the objective responses.

The clinical and translational findings from this study have the potential to inform rational decisions regarding combinations of treatment both in the metastatic and the adjuvant settings. This is a critical study to inform future practice and future phase 3 clinical trials. The translational research performed on tissue biopsies and blood will provide mechanistic information to guide the selection of optimal combinations of therapies for phase 3 studies in the advanced and the adjuvant setting.

This is a phase II, randomised, open label, three arm, parallel group, clinical trial of neoadjuvant combined targeted and immune therapy for patients with BRAF V600 mutant resectable stage III (bulky regional stage IIIB-D, but excluding in transit disease) melanoma.

This translational study explores pathological and RECIST response rates for a 6-week duration of neoadjuvant therapy across 3 treatment arms. The key secondary outcomes to be measured include a detailed analysis of immunologic, proteomic and genetic biomarkers in tumour tissue and peripheral blood at weeks 1, 2 and 6 compared to baseline and correlated with clinical, metabolic and pathological response to neoadjuvant treatment, and relapse and overall survival to adjuvant treatment. In patients who relapse within 40 weeks of adjuvant treatment, further analysis of tumour tissue (if possible) will be undertaken. Relapse free and overall survival, surgical outcomes and adverse event profile will also be determined.

Sixty patients will be randomised to one of three treatment groups in a 1:1:1 ratio, with 20 patients in each treatment arm:

* "Sequential immunotherapy": Dabrafenib 150mg orally twice a day + Trametinib 2mg orally once a day for 1 week, then followed by treatment with Pembrolizumab 2mg/kg delivered intravenously at weeks 1, 3, and 6, then once every 3 weeks from week 6 for 50 weeks.
* "Concurrent immunotherapy": Dabrafenib 150mg orally twice a day + Trametinib 2mg orally once a day + Pembrolizumab 200mg intravenously once every 3 weeks for 6 weeks then Pembrlizuamb alone for a further 46 weeks after surgery.
* "Immunotherapy alone": Pembrolizumab 200mg intravenously once every 3 weeks alone for 52 weeks.

Allocation of treatment will be concealed prior to randomisation which will be performed via a web based system in permuted blocks and stratified by BRAF V600E mutation versus non BRAF V600E mutation (i.e. V600D, V600K, V600R, V600M).

Neoadjuvant treatment for all three arms will be administered for 6 weeks, followed by complete resection of tumour to no evidence of disease. Surgery is followed by 46 weeks of pembrolizumab adjuvant therapy or until disease relapse, death, intolerable adverse drug reactions or by withdrawal of patient consent. After 52 weeks of the study treatment phase, patients will be followed 3 monthly for relapse (and progression, following relapse) and survival for 5 years.

The biomarker component of this study will require blood samples and core biopsies of tumour tissue at the following time points:

* Baseline (PRE)
* Week 1 (EDT 1)
* Week 2 (EDT 2)
* Week 6 - complete lymph node dissection specimen (POST)
* At Relapse (RELAPSE) if applicable and available

Surveillance of disease during the 6 week neoadjuvant period will be undertaken with surgical assessments and with ultrasounds of the affected lymph node basin.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Written informed consent.
* Histologically confirmed, resectable American Joint Committee on Cancer (AJCC, 8th edition) stage IIIB, IIIC (Tx, T0, T1-4, N1b, N2b, N3b, M0) cutaneous melanoma or unknown primary melanoma with sufficient cutaneous and/or nodal disease to enable multiple excisional or core biopsies (at baseline, week 1 and week 2). 'Resectable' tumours are defined as having no significant vascular, central nervous system or bony involvement. Only cases where a complete surgical resection with tumour-free margins can safely be achieved are defined as resectable. Patients who may not have sufficient disease to enable multiple biopsies at weeks 1 and 2 will not be excluded, however the intention of the study is that at least one biopsy at these time points is required.
* Measurable disease according to RECIST version 1.1 criteria (≥ 10mm longest diameter for non-nodal lesions and / or ≥ 15mm in shortest diameter for lymph nodes) within 4 weeks of randomisation. 'Measurable' disease may be ascertained by CT or for cutaneous and superficial lesions, by caliper measurement with digital photography. CT preferred for all lesions where possible. PET imaging will be performed, but not used for the primary purpose of measuring response.
* BRAF V600 mutation positive on immunohistochemistry or a local molecular test (e.g. Oncofocus): a. A positive V600E immunohistochemistry stain at study entry should be formally quantified with a local molecular test following study entry (e.g. Oncofocus); b. Molecular BRAF mutation status should preferentially be confirmed using tissue taken from the presenting stage III / IV disease. Alternatively, archival primary tissue is also acceptable to confirm BRAF mutation status.
* Able to swallow and retain oral medication
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Demonstrated adequate organ function as defined:

  1. Absolute neutrophil count (ANC) ≥1.5 109/L
  2. Platelets ≥100 109/L
  3. Haemoglobin ≥90g/L
  4. Serum creatinine OR measured or calculated creatinine clearance (CrCl) (Glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for patient with creatinine levels > 1.5 X institutional ULN.
  5. Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN.
  6. Aspartate transaminase (AST) and Alanine transaminase (ALT) ≤ 2.5 X ULN OR ≤ 5 X ULN for patients with liver metastases.
  7. Albumin >25 g/L
  8. International Normalized Ratio (INR) or Prothrombin Time (PT)
  9. Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants. ≤1.5 X ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Anticipated life expectancy of > 12 months.
* Women of childbearing potential: a negative serum pregnancy test within 72 hours of first dose of study treatment and effective contraception from 14 days prior to study treatment until 4 months after the last dose.
* Men with a female partner of childbearing potential to use effective contraception from 14 days prior to study treatment until 4 months after the last dose.

Exclusion Criteria:

* In transit disease
* Uveal or mucosal melanoma.
* Prior anti-cancer treatment for melanoma, except for the following:

  1. surgery for a primary melanoma or previous stage III melanoma,
  2. adjuvant radiotherapy to the primary melanoma resected site or to lymph nodes for previous Stage III disease,
  3. previous adjuvant interferon or ipilimumab for resected stage II or III melanoma, Previous adjuvant treatment with PD-1 inhibitors or BRAF/MEK inhibitors is not permitted.
* Received any investigational drug within 28 days or 5 half-lives of the planned first dose of this study treatment.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients and / or dimethyl sulfoxide (DMSO).
* Active infection requiring systemic therapy.
* Current use of any prohibited medication as described in protocol.
* Active autoimmune disease or a documented history of autoimmune disease or a syndrome requiring systemic steroids or immunosuppressive agents. Patients with the following are permitted to enrol:

  1. vitiligo,
  2. type I diabetes mellitus,
  3. residual hypothyroidism due to an autoimmune condition only requiring, and stable on hormone replacement,
  4. psoriasis not requiring systemic treatment,
  5. resolved childhood asthma or atopy,
  6. or conditions not expected to recur in the absence of an external trigger.
* A requirement for chronic systemic steroid therapy (> 10mg/kg per day of prednisone or equivalent) within two weeks before the planned first dose of study treatment or any on any other form of immunosuppressive treatment. Patients who require inhaled or intranasal corticosteroids (with minimal systemic absorption) may be continued if the patient is on a stable dose. Non-absorbed intra-articular steroid injections will also be permitted.
* A known history of another malignancy or concurrent malignancy unless the patient is disease-free for a minimum of 1 year, is completely treated and at low-risk of recurrence. The time requirement does not apply for patients with successful definitive resection or curative treatment of:

  1. Non-melanoma skin cancer (e.g. basal cell or squamous cell carcinoma of the skin),
  2. superficial bladder cancer,
  3. in situ carcinoma of the cervix,
  4. in situ breast cancer,
  5. atypical melanocytic hyperplasia or melanoma in situ
  6. other in situ carcinomas,
  7. multiple primary melanomas, or other treated low risk tumours.
* Known HIV, hepatitis B or C virus positive status or history of active tuberculosis (testing prior to randomisation is not required).
* Administration of a live vaccine with 30 days of planned first dose of study treatment. Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed, however intranasal influenza vaccines (e.g., Fluad®) are live attenuated vaccines, and are not allowed. Any vaccine is cautionary within 30 days.
* Patients with a history or evidence of cardiovascular risk including any of the following:

  1. QT interval corrected for heart rate using the Bazett formula ≥480 msec, a diagnosis of long QT syndrome (Roman-Ward or Jervell Lange-Nielsen syndromes)
  2. Taking medications known to prolong the QT interval.
  3. Uncorrectable electrolyte abnormal abnormality (e.g. hypo- or hyperkalaemia, hypomagnesaemia, hypocalcaemia)
  4. Uncontrolled arrhythmias, with the exception of atrial fibrillation which is controlled for > 30 days prior to randomisation.
  5. Patients with implanted cardioverter/defibrillators.
  6. Acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty or stenting within 6 months prior to randomisation.
  7. A history or current evidence of New York Heart Association (NYHA) ≥Grade 2 congestive heart failure
  8. A current left ventricular ejection fraction (LVEF) below than the lower limit of normal (LLN).
  9. Any abnormal cardiac valve morphology documented by echocardiogram which in the opinion of the investigator could interfere with the patient's safety.
  10. Treatment-refractory hypertension defined as a systolic blood pressure of >140 mm Hg and/or a diastolic pressure of >90 mm Hg, which cannot be controlled by anti-hypertensive treatment.
* Evidence or a risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR), including:

  1. Presence of predisposing factors to RVO or CSR (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled hypertension, uncontrolled diabetes mellitus, or a history of hyperviscosity or hypercoagulability syndromes).
  2. Visible retinal pathology as assessed by ophthalmic examination that is considered a risk factor for RVO or CSR, such as evidence of new optic disc cupping.
  3. Intraocular pressure > 21 mm Hg as measured by tonography.
  4. Evidence of new visual field defects on automated perimetry.
* History or evidence of interstitial lung disease or active non-infectious pneumonitis.
* Serious or unstable pre-existing medical conditions or other conditions that could interfere with the patient's safety, consent, or compliance.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or an agent directed to another co-inhibitory T-cell receptor (i.e. OX-40, CTLA-4).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2022-01-02 (Actual); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate | From baseline to 6 weeks
  Proportion of patients with complete absence of residual melanoma cells in the planned resected tumour site(s) at week 6 surgery.

SECONDARY OUTCOMES:
Objective clinical (RECIST) response rate | From baseline to 6 weeks
  Proportion of patients with complete and partial responses at 6 weeks compared to baseline per RECIST guidelines for each treatment arm.
Relapse free survival | 5 years
  The amount of time that patients are disease free from the time of surgery at 6 weeks from study entry
Overall survival | 5 years
  The proportion of patients who are alive from the time of study entry
Incidence of post operative infection | 6 weeks
  The number of patients (and the number of episodes) who develop a post operative infection of the surgical wound requiring intravenous antibiotics and/or wound drainage
Incidence of post operative seroma formation | 6 weeks
  The number of patients (and the number of episodes) who develop a seroma at the surgical site that requires any intervention and the volume of seroma drainage
Duration of post operative wound drainage time | 6 weeks
  The number of days that a wound drain remains in situ from the time of surgery
Incidence of post operative bleeding requiring return to theatre or transfusion | 6 weeks
  The number of patients (and the number of episodes) who have a bleed from the post operative surgical wound that requires a blood transfusion or return to theatre to stop the bleeding
Comparison of surgeon's opinion of operability evaluated at baseline to time of surgery | Baseline and 6 weeks
  The change, if any, in the surgeon's assessment of 'operability' from baseline opinion (based on clinical and imaging examination) to time of operation
Incidence of any treatment-emergent adverse events | 52 weeks
  The number of study treatment related adverse events of all Common Terminology Criteria for Adverse Events (CTCAE) grades from the time of starting study treatment to the time of permanent discontinuation of study treatment
Characterisation of the immunophenotype of tumour infiltrating cells in melanoma tissue | Baseline, Week 1, Week 2, Week 6
  The effects of study treatment on the body's immune cells within the tumour tissue prior to surgery
Description of the morphological assessment of melanoma tissue | Baseline, Week 1, Week 2, Week 6
  The effects of study treatment on the degree of necrosis and genetic markers in tumour tissue prior to surgery
Description of the RNA expression profile of melanoma tumour | Baseline, Week 1, Week 2, Week 6
  The effects of study treatment on the baseline function of RNA expression in tumour tissue prior to surgery
Measurement of leucocyte subpopulations in peripheral blood | Baseline, Week 1, Week 2, Week 6
  The effects of study treatment on the number and type of white cells in the blood
Measurement of circulating tumour DNA | Baseline, Week 1, Week 2, Week 6
  The levels of melanoma DNA that is circulating in the blood stream and the changes during study treatment

OTHER OUTCOMES:
Concordance of metabolic response measured by pathological response | 6 weeks
  The activity of melanoma tissue assessed by the uptake of fludeoxyglucose (18F) in tumour cells viewed using positron emission tomography (PET) and how well this corresponds to the findings from the pathological examination of completely excised tumour tissue
Concordance of metabolic response measured by RECIST response | 52 weeks
  The activity of melanoma tissue assessed by the uptake of fludeoxyglucose (18F) in tumour cells viewed using positron emission tomography (PET) and how well this corresponds to the assessment of tumour size and extent using computed tomography and magnetic resonance imaging scans
Concordance of pathological response measured by RECIST response | 6 weeks
  he findings from the pathological examination of completely excised tumour tissue and how well this corresponds to the assessment of tumour size and extent using computed tomography and magnetic resonance imaging scans
Concordance of metabolic response with RECIST response at relapse | 52 weeks
  The activity of recurrent melanoma tissue assessed by the uptake of fludeoxyglucose (18F) in tumour cells viewed using positron emission tomography (PET) and how well this corresponds to the assessment of tumour size and extent using computed tomography and magnetic resonance imaging scans
Concordance of immune related response criteria (irRC) with RECIST response | Weeks 6 and 52
  The application of two different criterion to establish the tumour burden as assessed with computed tomorgraphy and magnetic resonanse imaging
Correlation of the gut microbiome with RECIST response to immunotherapy. | Baseline, Week 6, week 24, at relapse if this occurs within 5 years from study entry
  Characterisation of the bacterial diversity and composition in stool samples at baseline, prior to surgery at week 6, week 24 and at relapse.
Characterisation of self-reported dietary habits (including use of oral probiotics) and correlation with the gut microbiome. | Baseline
  Diet plays a significant role in shaping the intestinal microbiome. Nutrition may influence the gut microbiome and response to immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Georgina V Long, Study Director — Melanoma Institute Australia
Locations (3):
- Australia (3):
  - Westmead Hospital, Sydney, New South Wales
  - Melanoma Institute Australia, Wollstonecraft, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Long GV, Carlino MS, Au-Yeung G, Spillane AJ, Shannon KF, Gyorki DE, Hsiao E, Kapoor R, Thompson JR, Batula I, Howle J, Ch'ng S, Gonzalez M, Saw RPM, Pennington TE, Lo SN, Scolyer RA, Menzies AM. Neoadjuvant pembrolizumab, dabrafenib and trametinib in BRAFV600-mutant resectable melanoma: the randomized phase 2 NeoTrio trial. Nat Med. 2024 Sep;30(9):2540-2548. doi: 10.1038/s41591-024-03077-5. Epub 2024 Jun 21. PMID 38907159
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215
- See also: Link to Registry Information on study of Neoadjuvant Dabrafenib + Trametinib for AJCC Stage IIIB-C BRAF V600 Mutation Positive Melanoma — https://clinicaltrials.gov/ct2/show/NCT01972347?term=neoadjuvant+melanoma+institute+australia&rank=1